CLINICAL TRIAL: NCT03749460
Title: Dual Immune Checkpoint Blockade and Hypofractionated Radiation in Patients With Salivary Gland Cancers
Brief Title: Nivolumab and Ipilimumab and Stereotactic Body Radiation Therapy in Treating Patients With Salivary Gland Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Cristina Rodriguez, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1718030; NCI-2018-02473 (Registry Identifier: NCI / CTRP); 8758 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Malignant Neoplasm in the Bone; Metastatic Malignant Neoplasm in the Lung; Salivary Gland Carcinoma; Stage IV Major Salivary Gland Cancer AJCC v8; Stage IVA Major Salivary Gland Cancer AJCC v8; Stage IVB Major Salivary Gland Cancer AJCC v8; Stage IVC Major Salivary Gland Cancer AJCC v8
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Nivolumab; Ipilimumab; CTLA-4 Antigen; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab, ipilimumab, SBRT) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 2 weeks for up to 12 courses and then every 4 weeks for an additional 8 courses in the absence of disease progression or unacceptable toxicity. Patients also receive ipilimumab IV over 60 minutes on day 1. Treatment repeats every 6 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity. Beginning week 3, patients undergo 3 fractions of stereotactic body radiation therapy every other day in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab; Biological: Ipilimumab; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Biological: Nivolumab — Given IV
  Other Names: 946414-94-4; BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo; CMAB819; Nivolumab Biosimilar CMAB819
Biological: Ipilimumab — Given IV
  Other Names: 477202-00-9; Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy; Biosimilar CS1002
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase I/II trial studies the side effects and how well nivolumab and ipilimumab works when given together with stereotactic body radiation therapy (SBRT) in treating patients with salivary gland cancers. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method can kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Giving nivolumab and ipilimumab and SBRT may work better in treating patients with advanced salivary gland cancers.

DETAILED DESCRIPTION:
Patients receive nivolumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 2 weeks for up to 12 courses and then every 4 weeks for additional 8 courses in the absence of disease progression or unacceptable toxicity. Patients also receive ipilimumab IV over 60 minutes on day 1. Treatment repeats every 6 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity. Beginning week 3, patients undergo 3 fractions of stereotactic body radiation therapy every other day in the absence of disease progression or unacceptable toxicity.

After completion of study treatment patients are followed up at 30 days and then every 8 or 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven salivary gland carcinoma (World Health Organization [WHO], 2005) arising from a previous head and neck primary site, and located within the head and neck region, lung or bone, and who are not candidates for curative intent therapy
* Demonstrated disease progression during, or after discontinuation, of the most recent line of systemic therapy. For patients who have received no prior systemic therapy, demonstrated progression in the 3 months prior to trial participation assessed by the treating physician
* Have received any number lines of prior systemic therapy (including systemic therapy in the curative intent setting)
* Have a lesion/s deemed suitable by the treating physicians for stereotactic body radiation therapy (SBRT) with the intent of palliation or prevention of symptoms. This lesion must be:

  * 1-3 non-overlapping sites in the head and neck region OR
  * Metastatic lesions outside the head and neck (H&N) region in the lung or bone (a minimum of 1 and a maximum 5 lesions will be irradiated), provided there is no significant overlap between the lesions ** Patients should have RECIST 1.1 criteria measurable disease in addition to the lesion/s treated with SBRT. If the site/s of SBRT were previously radiated to high dose radiation therapy (RT) (> 50Gy), there should be > 6 month time interval between the last dose of radiation and the start of SBRT
* Have the ability to tolerate required SBRT-related procedures (e.g.: lie flat and hold position for treatment) as determined by the treating physician
* Be willing and able to provide written informed consent for the trial and comply with the study visit requirements
* Have measurable disease based on RECIST 1.1. (in addition to the lesion/s that will be treated with stereotactic radiation therapy)
* Have provided tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion. Tissue requirement will be waived if deemed contraindicated or not clinically available/accessible for resection per the treating physician (principal investigator [PI] approval required)
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Hemoglobin >= 9.0 g/dL (performed within 28 days of treatment initiation)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9 /L (>= 1500 per mm^3) (performed within 28 days of treatment initiation)
* Platelet count >= 100 x 10^9 /L (>= 100,000 per mm^3) (performed within 28 days of treatment initiation)
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician (performed within 28 days of treatment initiation)
* Aspartate aminotransferases (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be =< 5 x ULN (performed within 28 days of treatment initiation)
* Serum creatinine clearance (CL) > 40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance (performed within 28 days of treatment initiation)
* Evidence of post-menopausal status OR negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy, or hysterectomy)
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)
* Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 1 method of highly effective birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 180 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 180 days after the last dose of study therapy
* Patient is >= 5 years free of another primary malignancy, except:

  * If the other malignancy is basal cell carcinoma or cervical carcinoma in situ or
  * If the other primary malignancy is not considered clinically significant and is requiring no active intervention

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment
* Has a target lesion/s for SBRT that demonstrate any of the following:

  * Located within 2 cm of the proximal bronchial tree
  * > 5 cm (> 50 cc) in greatest dimension
* Has a target lesion/s in a region that previously received high dose radiation therapy (RT) (> 50 Gy) demonstrating any of the following:

  * Carotid artery encasement (> 180 degrees) (due to risk of carotid blow out)
  * Unprotected carotid artery (i.e. skin is directly over the carotid without intervening soft tissue, especially after prior neck dissection without a vascularized free flap) (due to risk of carotid blow out)
  * Skin infiltration by tumor (due to risk of fistula)
  * Located in the larynx/hypopharynx primaries (due airway threat)
  * Treated with high dose radiation therapy (> 50 Gy) within 6 months or less of trial enrollment
* Prior receipt of an anti-PD-1, anti-PDL1 or anti-CTLA4 immune checkpoint inhibitor
* Current or prior use of immunosuppressive medication within 14 days before the first dose of nivolumab or ipilimumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication)
* Has received a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., =< Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has received prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., =< Grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Subjects with =< Grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Has known brain metastases or spinal cord compression unless the patient is stable (asymptomatic; no evidence of new or emerging brain metastases; and stable and off steroids for at least 14 days prior to start of study treatment). Following radiotherapy and/or surgery of the brain metastases patients must wait 4 weeks following the intervention and before initiating study treatment with imaging to confirm stability
* Has an active autoimmune disease requiring systemic treatment within the past 2 years or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement will not be excluded from the study
* Has a history of or evidence of active interstitial lung disease or non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 180 days after the last dose of trial treatment
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has evidence of acute or chronic hepatitis B, or hepatitis C
* Has received a live vaccine within 30 days prior to the first dose of trial treatment
* Has a history of primary immunodeficiency or an allogeneic organ transplant
* Known history of previous clinical diagnosis of tuberculosis
* Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2023-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Rodriguez, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Nivolumab, Ipilimumab, SBRT)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nivolumab, Ipilimumab, SBRT)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: Years] | 56.4 [27 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Toxicity Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0
Description: Toxicities will be summarized as the number and percentage of patients with each type of toxicity, per Criteria for Adverse Events version 5.0
Time Frame: From start of treatment through up to 100 days after the completion of study treatment (up to 16 months total)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nivolumab, Ipilimumab, SBRT)
Number analyzed (Participants) | 20
Participants
  Adrenal Insufficiency | 3
  Allergic Reaction | 1
  Anemia | 2
  Anorexia | 6
  Anxiety | 2
  Arthralgia | 2
  Arthritis | 2
  Aspirational Pneumonitis | 1
  Hyperthyroidism | 1
  Back Pain | 2
  Bilateral Upper Extremity Edema | 1
  Non-Cardiac Chest Pain | 3
  Chills | 1
  Confusion | 1
  Congestion | 1
  Conjuctival Erythema | 1
  Constipation | 7
  Cough | 5
  Dehydration | 1
  Depression | 1
  Diarrhea | 5
  Dysphagia | 1
  Drooling | 1
  Dry Eyes | 3
  Dry Mouth | 3
  Dry Skin | 2
  Dyspnea | 4
  Ear Fullness | 1
  Alkaline Phophate Increased | 1
  Asparate Aminotransferase Increased | 1
  Alanine Aminotransferase Increased | 1
  Epistaxis | 3
  Esophagitis | 1
  Fall | 1
  Fatigue | 15
  Erythematous Pustular Rash | 1
  Fistual Tract | 1
  Flu Like Symptoms | 1
  Fungal Infection | 1
  GERD | 2
  Hair Loss | 1
  Hallucinations | 1
  Head/Neck Swelling | 1
  Headache | 4
  Hearing Loss | 1
  Heartburn | 2
  Hemoptysis | 1
  Hot Flashes | 1
  Hyperpigmented Skin | 1
  Hypertension | 2
  Hypoalbuminemia | 1
  Hypocalcemia | 1
  Hypothyroidism | 5
  Increased Spine Pain | 1
  Worsening Trismus | 1
  Swollen Neck Sore | 1
  Hypokalemia | 3
  Infusion Related Reaction | 5
  Insomnia | 6
  Intermittent Palpatations | 1
  Intermittent Abdominal Cramping | 1
  Intermittent Dizziness | 3
  Intermittent Facial Swelling | 1
  Intermittent Hypertension | 1
  Intermittent Maculopapular rash | 1
  Intermittent Nasal Congestion | 1
  Intermittent Rhinitis | 1
  Joint Pain | 1
  Ear Bleeding | 1
  Facial Neuropathy | 1
  Left Neck Discomfort | 1
  Neck Pain | 2
  Lower Extremity Edema | 1
  Lung Infection (Pneumonia) | 2
  Lymphedema | 1
  Maculopapular Rash | 4
  Mania | 1
  Mental Fogginess | 1
  Microcytic Anemia | 1
  Mucositis | 5
  Pustular Skin Rash | 1
  Muscle Weakness | 1
  Muscle Spams | 1
  Myalgias | 4
  Nausea | 10
  Neck Tightness | 1
  Neuropathy | 1
  Night Sweats | 1
  Non Pruritic Cheek Rash | 1
  Otorrhea | 1
  Skin Pain | 1
  Facial Pain | 1
  Pruritus | 5
  Rash | 1
  Renal Insufficiency | 1
  Respiratory Infection | 1
  Itchy Eyes | 1
  Eye Pain | 1
  Foot Pain | 1
  Right Knee Fracture | 1
  Foot Edema | 1
  Periorbital Edema | 1
  Thoracic Pain | 1
  Rhinorrhea | 2
  Cancer Related Pain | 1
  Right Leg Pain | 1
  Sinus Congestion | 2
  Skin Infection | 1
  Sore Throat | 2
  Hyperhidrosis | 1
  Swollen Joints | 1
  Taste Changes | 3
  Upper Respiratory Infection | 2
  Urinary Frequency | 1
  Urinary Tract Infection | 1
  Vision Changes | 2
  Vomiting | 1
  Abdominal Pain | 4
  Weight Loss | 4
  Hoarseness | 1
  Tinnitus | 1
  Xerostomia | 1
  Dyspepsia | 1
  Right Rib Fracture | 1
  Right Coracoid Fracture | 1
  Oral Bleeding | 1
  Hypotension | 1

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Clinical responses to the combination of nivolumab, ipilimumab and hypofractionated radiation will be based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nivolumab, Ipilimumab, SBRT)
Number analyzed (Participants) | 20
Participants
  Stable Disease | 6
  Progressive Disease | 10
  Partial Response | 4

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS estimate will be calculated using the Kaplan-Meier method. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesion
Time Frame: From the date of study enrollment, until disease progression or death, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Nivolumab, Ipilimumab, SBRT)
Number analyzed (Participants) | 20
Months | 7.2 [2.52 to 18.24]

4. Secondary Outcome: Overall Survival (OS)
Description: OS estimate will be calculated using the Kaplan-Meier method.
Time Frame: From the date of study enrollment, until disease progression or death, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Nivolumab, Ipilimumab, SBRT)
Number analyzed (Participants) | 20
months | 25 [18.72 to 31.08]

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: Adverse events are collected from the first dose of Ipilimumab/Nivolumab, and are collected through 100 days post the last dose of therapy.
Arm/Group | Treatment (Nivolumab, Ipilimumab, SBRT)
All-Cause Mortality (participants affected / at risk) | 9/20
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nivolumab, Ipilimumab, SBRT) (N=20)
Right Rib Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Right Coracoid Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 1 (1)
Oral Bleeding (General disorders) | 1 (1)
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pneumonia
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nivolumab, Ipilimumab, SBRT) (N=20)
Abdominal Pain (Gastrointestinal disorders) | 4 (7)
Adrenal Insufficiency (Endocrine disorders) | 3 (3)
Allergic Reaction (Immune system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Anxiety (Psychiatric disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Aspirational Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bilateral Upper Extremity Edema (General disorders) | 1 (1)
Non-Cardiac Chest Pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Chills (General disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Conjuctival Erythema (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Drooling (Nervous system disorders) | 1 (1)
Dry Eyes (Eye disorders) | 3 (3)
Dry Mouth (Gastrointestinal disorders) | 3 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Ear Fullness (Ear and labyrinth disorders) | 1 (1)
Alkaline Phosphate Increased (Investigations) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 15 (16)
Erythematous-Pustular Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Fistula Tract (Skin and subcutaneous tissue disorders) | 1 (1)
Flu Like Symptoms (General disorders) | 1 (1)
Fungal Infection (Infections and infestations) | 1 (1)
GERD (Gastrointestinal disorders) | 2 (2)
Hair Loss (Skin and subcutaneous tissue disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Head/Neck Swelling (General disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Hearing Loss (Ear and labyrinth disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 2 (2)
Hemoptysis (Gastrointestinal disorders) | 1 (1)
Hot Flashes (General disorders) | 1 (1)
Hyperpigmented Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (4)
Hypoalbuminemia (Blood and lymphatic system disorders) | 1 (1)
hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 5 (5)
Increased Spine Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Worsening Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Swollen Neck Sore (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 5 (7)
Insomnia (Psychiatric disorders) | 6 (6)
Intermittent Palpitations (Cardiac disorders) | 1 (1)
Intermittent Abdominal Cramping (Gastrointestinal disorders) | 1 (1)
Intermittent Dizziness (Nervous system disorders) | 2 (2)
Intermittent Facial Swelling (General disorders) | 1 (1)
Intermittent Hypertension (Cardiac disorders) | 1 (1)
Intermittent Maculopapular Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Intermittent Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intermittent Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Ear Bleeding (Ear and labyrinth disorders) | 1 (1)
Facial Neuropathy (Nervous system disorders) | 1 (1)
Left Neck Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Lower Extremity Edema (Vascular disorders) | 1 (1)
Lung Infection (Pneumonia) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1)
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Mania (Psychiatric disorders) | 1 (1)
Mental Fogginess (Nervous system disorders) | 1 (1)
Microcytic Anemia (Blood and lymphatic system disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 5 (6)
Pustular Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgias (Musculoskeletal and connective tissue disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 10 (13)
Neck Tightness (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Night Sweats (General disorders) | 1 (1)
Non Pruritic Cheek Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Otorrhea (Ear and labyrinth disorders) | 1 (1)
Skin Pain (Skin and subcutaneous tissue disorders) | 1 (1)
Facial Pain (General disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Renal Insufficiency (Renal and urinary disorders) | 1 (1)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Itchy Eyes (Eye disorders) | 1 (1)
Eye Pain (Eye disorders) | 1 (1)
Foot Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Right Knee Fracture (Injury, poisoning and procedural complications) | 1 (1)
Foot Edema (General disorders) | 1 (1)
Periorbital Edema (General disorders) | 1 (1)
Thoracic Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cancer Related Pain (Gastrointestinal disorders) | 1 (2)
Right Leg Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Skin Infection (Skin and subcutaneous tissue disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Swollen Joints (Musculoskeletal and connective tissue disorders) | 1 (1)
Taste Changes (Gastrointestinal disorders) | 3 (3)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Urinary Frequency (Renal and urinary disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Vision Changes (Eye disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight Loss (Metabolism and nutrition disorders) | 4 (4)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Xerostomia (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT03749460/Prot_SAP_000.pdf